CLINICAL TRIAL: NCT00177801
Title: Organ Transplant Infection Prevention and Detection Project 1.0; Cohort Study of Transplant Recipients at "Ultra-High" Risk for Invasive Fungal Infections
Brief Title: Organ Transplant Infection Prevention and Detection Project
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB# 0408132; CDC
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Transplantation Infection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. The biologic samples may be given to the Centers for Disease Control and Prevention. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fungal infections are leading causes of morbidity and mortality in transplant recipients, yet comprehensive epidemiologic studies in this area are lacking. For this reason, the Centers for Disease Control and Prevention have provided a grant to the University of Pittsburgh to study this subject.

The study has four specific aims:

1. To determine the risk of fungal infections in a center where "tolerogenic" immunosuppressive protocols are currently in place, and to determine whether there are any measures of immune system function which correlate with risk of fungal infection.

2: To create a repository of serum, urine and bronchoalveolar lavage specimens for the purpose of determining the effectiveness of novel diagnostic tests for invasive fungal infections. Such a repository could also be utilized for the purpose of determining the effectiveness of novel diagnostic tests for viral infections such as West Nile Virus, cytomegalovirus, HHV-6 and HHV-8.

Specific aim 1 will be investigated by creating a prospective database of solid organ transplant recipients at the University of Pittsburgh Medical Center, including demographic factors as well as subsequent development of infection. The immune function of patients will be assessed by measuring T cell subsets and assessing T cell function using the Cylex assay. Specific aim 2 involves collection of serum, urine and bronchoalveolar lavage fluid. These specimens will be stored and later tested at the Centers for Disease Control and Prevention in the assessment of novel tests developed for the diagnosis of invasive fungal infections.

DETAILED DESCRIPTION:
This is a longitudinal cohort study. Participation in the research database is limited to placement of the subjects' identifiable medical information related to their organ transplantation and immunosuppression use. Participants can consent to allow only medical information collected and/or provide blood and tissue samples.

Patients seen by the Infectious Disease/Transplant team will be asked to provide their written informed consent to allow their past, current and future identifiable medical record information related to their condition placed in the research database. The medical record information that will be placed in the database will be related directly to the patients'-participants' disease process. However, since concurrent medical conditions and treatments (i.e., not related directly to transplantation) may impact substantially the patients'-participants' condition, it is likely that all of the patients'-participants' past, current and future identifiable medical record information will be placed in the research database. Consent will be obtained in the pre-transplant period. The advantage of this system is that consent is obtained directly from the patient (rather than from a proxy, as would be necessary in situations where consent is obtained post-transplant). Secondly, since the timing transplantation can not be predicted with certainty and may occur at hours during which research coordinators are not working, consent prior to transplantation ensures that the entire post-transplant period is covered by consent. This would ensure that early post-transplant infections are not missed, thereby eliminating a form of systematic bias. The disadvantage of this system is that some patients undergo informed consent who do not subsequently undergo transplantation. Additionally, occasional patients who present with acute organ system failure (for example, patients with fulminant hepatic failure) will not undergo pre-transplant consent. We will attempt to minimize this risk by pre-study and subsequent meetings with transplant surgeons to ensure the study team is informed about such patients on a timely basis.

Participant medical information will be stored electronically within the research data base.

The names, social security numbers, and medical record numbers of the participants will be deleted from their stored medical information and replaced with a linkage code. Access to participant medical information contained within the research database will be restricted to the research investigator and research staff..

Information linking the linkage codes to the participants' names, social security numbers and medical record numbers will be stored in a secure location separate from the medical information. Access to the information linking the linkage codes with participant names, social security numbers and medical record numbers will be granted only to the Principal Investigator and research coordinator of this research database.

Participant medical record information will be stored in the research database for an indefinite period of time.

The participant will be followed for up to four years after transplantation.

Epidemiologic information to be collected

At baseline (upon signing informed consent), the following information will be collected: Demographic data - age, sex, state of birth, prior travel to an area endemic for histoplasmosis, coccidioidomycosis or blastomycosis, indication for listing for transplantation, other prior medical problems, prior chemotherapy/immunosuppressive therapies and prior fungal infections.

During the first week post transplant, the following information will be collected: Type and date of transplant, UNOS status, pre-transplant conditioning with thymoglobulin or alemtuzumab, ongoing immunosuppressive regimen. At the time of fungal infection, the following information will be collected - symptoms and signs of infection and their duration, receipt of antifungal prophylaxis, presence of indwelling vascular devices, duration of neutropenia, presence of graft versus host disease (GVHD) and its severity and treatment, history of graft rejection and its treatment

Six weeks following the fungal infection, the following information will be collected - treatment of the infection, outcome (including duration of hospitalization, fate of organ graft and mortality)

Blood work to be collected

A separate consent form will be presented for blood work. This is to ensure that the patients who decline blood work specifically for the study still have the opportunity to have their epidemiologic information collected. The following tests will be collected specifically for the study.

* CD4 lymphocyte count pre-transplant and then every three months post-transplant
* Blood for Cylex assay pre-transplant then once per month X18 months
* Blood for storage (see below)* Additionally, bronchoalveolar lavage fluid will be collected (see below for schedule)

  *Blood for storage will be collected on those patients at highest risk for invasive fungal infections (4, 11, 42, 43). These patients will be:
* Lung transplant recipients
* Intestinal transplant recipients
* Kidney/pancreas transplant recipients
* Liver transplant recipients on renal replacement therapy or requiring re-transplantation in the first week post-transplantation

The BAL samples will be collected only if the subject undergoes a clinically indicated bronchoscopy and only the excess BAL fluid will be collected for the study.

Mycologic samples

All fungi grown from routine clinical specimens from patients in the study will be saved by the clinical microbiology laboratory. They will be made available to the Centers for Disease Control and Prevention (CDC) - other researchers working in conjunction with the CDC may also examine these isolates for mechanisms of antifungal resistance or mechanisms of pathogenicity. No patient identifiers would be provided to either the CDC or to other researchers. Only relevant "de-identified" clinical information (eg, prior use of specific antifungal agents) would be provided.

ELIGIBILITY:
Inclusion Criteria:

* will to sign consent
* speak English
* On lung transplant list awaiting lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplant recepients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pitttsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States